CLINICAL TRIAL: NCT06361927
Title: A Phase II Study of SSGJ-707 Monotherapy in First-line PD-L1 Positive Advanced NSCLC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-707-NSCLC-II-01
Record Dates: First submitted 2024-04-08; First posted 2024-04-12 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- cohort A：dose level 1 of SSGJ-707 (Experimental)
  Interventions: Drug: SSGJ-707
- cohort A：dose level 2 of SSGJ-707 (Experimental)
  Interventions: Drug: SSGJ-707
- cohort A：dose level 3 of SSGJ-707 (Experimental)
  Interventions: Drug: SSGJ-707
- cohort B：dose level 1 of SSGJ-707 (Experimental)
  Interventions: Drug: SSGJ-707
- cohort B：dose level 2 of SSGJ-707 (Experimental): cohort B
  Interventions: Drug: SSGJ-707
- cohort B：dose level 3 of SSGJ-707 (Experimental)
  Interventions: Drug: SSGJ-707

INTERVENTIONS:
Drug: SSGJ-707 — bispecific antibody

SUMMARY:
This study includes two cohorts, cohort A is for non-squamous NSCLC and cohort B is for squamous NSCLC.

DETAILED DESCRIPTION:
This study is a study of SSGJ-707 monotherapy in First-line PD-L1 Positive advanced NSCLC Patients. This study includes two cohorts, cohort A is for non-squamous NSCLC and cohort B is for squamous NSCLC. Each cohort will assess the efficacy and safety of the preset several dose levels of SSGJ-707 in advanced NSCLC Patients.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females over age 18
2. Histologically and/or cytologically documented local advanced or metastatic NSCLC .
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
4. Expected survival >=3 months.
5. Signed informed consent form.

Exclusion Criteria:

1. Known uncontrolled or symptomatic central nervous system metastatic disease.
2. Adverse events (with exception of alopecia and fatigue) from any prior anticancer therapy of grade >1 (National Cancer Institute Common terminology Criteria [NCI CTCAE] v.5.0).
3. Inadequate organ or bone marrow function.
4. Pregnant or breast-feeding woman.
5. Known allergies, hypersensitivity, or intolerance to SSGJ-707. The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 months
  Objective response rate

SECONDARY OUTCOMES:
Safety and tolerability | 12 months
  Safety and tolerability assessed by incidence and severity of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Lin Wu, MD, Ph.D, Principal Investigator — The Hunan Cancer Hospital
Locations (1):
- The Hunan Cancer Hospital, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No